CLINICAL TRIAL: NCT04548219
Title: Relative Bioavailability of a Mirikizumab Test Formulation Compared to the Reference Formulation in Healthy Subjects
Brief Title: A Study to Compare Two Different Formulations of Mirikizumab in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17667; I6T-MC-AMBV (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-09-10; First posted 2020-09-14 (Actual); Results first posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2023-05

CONDITIONS: Healthy
MeSH Terms: interventions — mirikizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mirikizumab (Reference) (Experimental): 200 milligram (mg) of mirikizumab as reference formulation (100 mg/mL), 2 × 1-mL pre-filled syringe administered as a subcutaneous (SC) injection into the arm/thigh/abdomen on day 1.
  Interventions: Drug: Mirikizumab
- Mirikizumab (Test) (Experimental): 200 mg of mirikizumab as test formulation (100 mg/mL), 2 × 1-mL pre-filled syringe administered as a SC injection into the arm/thigh/abdomen on day 1.
  Interventions: Drug: Mirikizumab

INTERVENTIONS:
Drug: Mirikizumab — Reference and test formulations of mirikizumab administered as a SC injection.
  Other Names: LY3074828

SUMMARY:
The purpose of this study is to compare two different formulations of mirikizumab in healthy participants. This study will compare how much of each formulation gets into the blood stream and how long it takes the body to remove it. Information about any side effects that may occur will also be collected. Participants will remain in the study for about 12 weeks, after receiving study drug.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or females, as determined through medical history and physical examination

Exclusion Criteria:

* Must not have an average weekly alcohol intake that exceeds 21 units/week (males) and 14 units/week (females)
* Must not show evidence of active or latent tuberculosis (TB)
* Must not have received live vaccine(s) (including attenuated live vaccines and those administered intranasally) within 8 weeks of screening, or intend to during the study
* Must not have been treated with steroids within 1 month of screening, or intend to during the study
* Must not be immunocompromised
* Must not have received treatment with biologic agents (e.g. monoclonal antibodies, including marketed drugs) within 3 months or 5 half-lives (whichever is longer) prior to Day 1
* Must not have clinically significant multiple or severe drug allergies, or intolerance to topical corticosteroids, or severe post treatment hypersensitivity reactions
* Must not have had lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years
* Must not have had breast cancer within the past 10 years
* Must not have significant allergies to humanized monoclonal antibodies
* Must not have clinically significant multiple or severe drug allergies, or intolerance to topical corticosteroids, or severe post treatment hypersensitivity reactions

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2021-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- QPS, Springfield, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Otani Y, Feagan BG, D'Haens GR, Escobar R, Morris NJ, Payne CD, Ugolini Lopes M, Zhang X. Pharmacokinetic Comparability and Safety Between Original and Citrate-Free Mirikizumab Formulations for Subcutaneous Injections: Results from Three Clinical Trials. Adv Ther. 2025 May;42(5):2369-2384. doi: 10.1007/s12325-025-03158-y. Epub 2025 Mar 21. PMID 40117091

RESULTS

PARTICIPANT FLOW:
Groups:
- 200 Milligram (mg) Mirikizumab (Reference): Arm: Participants received 200 mg mirikizumab reference formulation (100 mg/mL), 2 × 1-mL pre-filled syringe administered as a subcutaneous (SC) injection into the arm on day 1.
- 200 mg Mirikizumab (Reference): Thigh: Participants received 200 mg mirikizumab reference formulation (100 mg/mL), 2 × 1-mL pre-filled syringe administered as a SC injection into the thigh on day 1.
- 200 mg Mirikizumab (Reference): Abdomen: Participants received 200 mg mirikizumab reference formulation (100 mg/mL), 2 × 1-mL pre-filled syringe administered as a SC injection into the abdomen on day 1.
- 200 mg Mirikizumab (Test): Arm: Participants received 200 mg mirikizumab test formulation (100 mg/mL), 2 × 1-mL pre-filled syringe administered as a SC injection into the arm on day 1.
- 200 mg Mirikizumab (Test): Thigh: Participants received 200 mg mirikizumab test formulation (100 mg/mL), 2 × 1-mL pre-filled syringe administered as a SC injection into the thigh on day 1.
- 200 mg Mirikizumab (Test): Abdomen: Participants received 200 mg mirikizumab test formulation (100 mg/mL), 2 × 1-mL pre-filled syringe administered as a SC injection into the abdomen on day 1.
Period: Overall Study
Arm/Group | 200 Milligram (mg) Mirikizumab (Reference): Arm | 200 mg Mirikizumab (Reference): Thigh | 200 mg Mirikizumab (Reference): Abdomen | 200 mg Mirikizumab (Test): Arm | 200 mg Mirikizumab (Test): Thigh | 200 mg Mirikizumab (Test): Abdomen
Started | 10 | 10 | 10 | 10 | 10 | 10
Received at Least 1 Dose of Study Drug | 10 | 10 | 10 | 10 | 10 | 10
Completed | 10 | 10 | 10 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- 200 mg Mirikizumab (Reference): Participants received 200 mg mirikizumab reference formulation (100 mg/mL), 2 × 1-mL pre-filled syringe administered as a SC injection into the arm/thigh/abdomen on day 1.
- 200 mg Mirikizumab (Test): Participants received 200 mg mirikizumab test formulation (100 mg/mL), 2 × 1-mL pre-filled syringe administered as a SC injection into the arm/thigh/abdomen on day 1.
- Total: Total of all reporting groups
Arm/Group | 200 mg Mirikizumab (Reference) | 200 mg Mirikizumab (Test) | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 27 | 53
  >=65 years | 4 | 3 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 22 | 41
  Male | 11 | 8 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 30 | 29 | 59
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 29 | 29 | 58
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Mirikizumab
Description: PK: Cmax of mirikizumab was evaluated.
Time Frame: Predose on Day 1, Day 3, Day 5, Day 8, Day 11, Day 15, Day 22, Day 29, Day 43, Day 57, Day 71 and Day 85 postdose
Population: All participants who received at least 1 dose of study drug (mirikizumab) and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (ug/mL)
Arm/Group | 200 mg Mirikizumab (Reference) | 200 mg Mirikizumab (Test)
Number analyzed (Participants) | 30 | 30
micrograms per milliliter (ug/mL) | 12.7 (48) | 11.6 (45)
Statistical Analysis 1: Comparison: 200 mg Mirikizumab (Reference) vs 200 mg Mirikizumab (Test); Test type: Other — A linear fixed-effects model is used to estimate the relative bioavailability; Ratio of Geometric least squares mean = 0.907, 90% CI 2-sided [0.775 to 1.06]

2. Primary Outcome: PK: Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC[0-inf]) of Mirikizumab
Description: PK: AUC(0-inf) of mirikizumab was evaluated.
Time Frame: Predose on Day 1, Day 3, Day 5, Day 8, Day 11, Day 15, Day 22, Day 29, Day 43, Day 57, Day 71 and Day 85 postdose
Population: All participants who received at least 1 dose of study drug (mirikizumab) and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*day/mL
Arm/Group | 200 mg Mirikizumab (Reference) | 200 mg Mirikizumab (Test)
Number analyzed (Participants) | 30 | 30
ug*day/mL | 229 (56) | 209 (45)
Statistical Analysis 1: Comparison: 200 mg Mirikizumab (Reference) vs 200 mg Mirikizumab (Test); Test type: Other — A linear fixed-effects model is used to estimate the relative bioavailability; Ratio of Geometric least squares mean = 0.915, 90% CI 2-sided [0.761 to 1.10]

3. Primary Outcome: PK: Area Under the Concentration Versus Time Curve From Time Zero to t, Where t is the Last Timepoint With a Measurable Concentration (AUC[0-tlast]) of Mirikizumab
Description: PK: (AUC[0-tlast]) of mirikizumab was evaluated.
Time Frame: Predose on Day 1, Day 3, Day 5, Day 8, Day 11, Day 15, Day 22, Day 29, Day 43, Day 57, Day 71 and Day 85 postdose
Population: All participants who received at least 1 dose of study drug (mirikizumab) and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*day/mL
Arm/Group | 200 mg Mirikizumab (Reference) | 200 mg Mirikizumab (Test)
Number analyzed (Participants) | 30 | 30
ug*day/mL | 225 (56) | 206 (46)
Statistical Analysis 1: Comparison: 200 mg Mirikizumab (Reference) vs 200 mg Mirikizumab (Test); Test type: Other — A linear fixed-effects model is used to estimate the relative bioavailability; Ratio of Geometric least squares mean = 0.915, 90% CI 2-sided [0.760 to 1.10]

ADVERSE EVENTS:
Time Frame: Up To 85 Days
Description: All participants who received at least 1 dose of study drug.
Groups:
- 200 mg Mirikizumab (Reference): Arm: Participants received 200 mg mirikizumab reference formulation (100 mg/mL), 2 × 1-mL pre-filled syringe administered as a SC injection into the arm on day 1.
Arm/Group | 200 mg Mirikizumab (Reference): Arm | 200 mg Mirikizumab (Reference): Thigh | 200 mg Mirikizumab (Reference): Abdomen | 200 mg Mirikizumab (Test): Arm | 200 mg Mirikizumab (Test): Thigh | 200 mg Mirikizumab (Test): Abdomen
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 2/10 | 1/10 | 0/10 | 0/10 | 3/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 200 mg Mirikizumab (Reference): Arm (N=10) | 200 mg Mirikizumab (Reference): Thigh (N=10) | 200 mg Mirikizumab (Reference): Abdomen (N=10) | 200 mg Mirikizumab (Test): Arm (N=10) | 200 mg Mirikizumab (Test): Thigh (N=10) | 200 mg Mirikizumab (Test): Abdomen (N=10)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anosmia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-08-17): https://cdn.clinicaltrials.gov/large-docs/19/NCT04548219/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-18): https://cdn.clinicaltrials.gov/large-docs/19/NCT04548219/SAP_001.pdf